CLINICAL TRIAL: NCT04750109
Title: Carcinoma of Unknown Primary (CUP): a Comparison Across Tissue and Liquid
Brief Title: Carcinoma of Unknown Primary (CUP): a Comparison Across Tissue and Liquid Biomarkers
Acronym: CUP-COMP
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Hoffmann-La Roche (Industry); Concr (Industry); Durham University (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp188
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples will be collected for translational research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients with Carcinoma of Unknown Primary (CUP) have widespread cancer at diagnosis however the specific site of origin cannot be found, despite significant testing, making it difficult to treat. CUP has a poor prognosis; it is the 6th most common cause of cancer death in the UK.

To date there have been limited studies investigating molecular genomics in CUP patients, resulting in limited evidence to evaluate whether genomic profiling has added value over and above the standard diagnostics provided in the NHS.

As a result, our project will aim to;

* Assess genomic sequencing (both in tissue and blood) for the diagnosis and treatment guidance in CUP patients including a comparison of the effectiveness of tissue and blood based biomarkers
* Collect evidence to further develop technology that predicts an individual's response to a treatment
* Develop innovative systems of clinical data capture in patients with CUP
* Investigate novel biomarkers to determine the primary tumour location Approximately 120-140 CUP patients will be recruited across 7 UK NHS sites. Tumour samples will be collected from patients undergoing a standard of care procedure OR medically fit patients with accessible tumour. Archival tumour may also be obtained. Some samples will be stored for future translational research.

Sequencing results alongside clinical data will be discussed by a multi-disciplinary CUP Molecular Tumour Board. They will provide oversight on the nature, clinical significance and relevance of the results. They will inform the local CUP team of any "actionable" genetic changes, which could potentially direct selection of a targeted therapy trial for that patient. Sequential blood samples will be collected to investigate genetic characteristics that may be able to predict response to therapy.

The aggregated anonymised data will be made publicly available following completion of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or over
* Written informed consent according to ICH/GCP and national regulations
* ECOG Performance status 0-2
* Confirmed diagnosis of CUP as per the ESMO guidelines (described above). Patients must have;

  1. The local pathology reports confirming compatibility with CUP diagnosis and the associated slides used for the diagnosis
  2. Discussion at a local CUP MDT confirming diagnosis
* Accessible tumour that can be safely biopsied using radiological techniques. Biopsy may be undertaken as standard of care (surplus tissue sample to be used for this protocol), or maximum of one fresh biopsy specifically for purposes of the protocol. Subjects with inaccessible tumours for biopsy specimens but with a confirmed CUP diagnosis, may be enrolled without a biopsy upon consultation and agreement by the sponsor
* Availability of archival tumour sample, slides and histological report
* Willingness to provide blood samples on up to three occasions during the course of the study

Exclusion Criteria:

* Patient with an immunohistochemistry profile that provides a definitive clinical indication of a primary cancer with a specific treatment
* Known HIV, Hepatitis B, C positive, or COVID-19 positive, due to the difficulties in handling high-risk specimens
* Patients who are unable to provide fully informed written consent
* Presence of any medical, psychological, familial or sociological condition that, in the investigator's opinion, will hamper compliance with the study protocol and follow-up schedule
* Bleeding diathesis (patients' on anticoagulation are permitted to enter the trial if anticoagulation can be safely managed to enable fresh tumour biopsies and blood sampling)
* Conditions in which research biopsies or blood sampling may increase risk of complications for the patients and/or investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All study participants must have a histological confirmed diagnosis of CUP based on the clinical, radiological and pathological review at a local or regional CUP MDT and the 2015 ESMO Clinical Practice Guidelines for CUP(Fizazi et al., 2015). Favourable and unfavourable-risk CUP subsets are eligible. The population to be included in this study corresponds to patients with CUP of epithelial origin for whom a likely tissue of origin cannot be determined.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
To sequence tumour tissue and circulating tumour DNA from approximately 120- 140 patients with CUP in order to evaluate the activation state of various oncogenic pathways and improve treatment stratification approaches | 18 months
To establish a genomic reporting mechanism whereby clinically relevant and potentially 'actionable' abnormalities found during sequencing/molecular characterisation can be reported to patients | 18 months

SECONDARY OUTCOMES:
To obtain archival tumour specimens, fresh tissue and sequential blood samples from approximately 120 - 140 patients with CUP | 18 months
The comparative assessment of alternative assay methods (such as ctDNA) in parallel with whole genome sequencing in the diagnosis and treatment stratification for patients with CUP | 18 months
To collect samples for future analysis for additional molecular characterisation techniques for detection of actionable aberrations. Examples include RNA sequencing, IHC, proteomics, methylation, analysis of immuno-biomarkers | 18 months
To perform whole genome sequencing in patients where enough tumour tissue is available to explore novel predictive and resistance biomarkers | 18 months
To build on close collaborations between the NHS CUP Hospitals, and external collaborators to progress basic/translational research models to investigate biomarkers to treatment in CUP and key biological drivers of this disease. | 18 months
Collect evidence investigating the most effective way to stratify patients with CUP onto treatment. | 18 months
To understand whether liquid biomarkers in CUP can be used to stratify patients and give prognostic information | 18 months
Develop a data collection repository within the NHS for patients with CUP | 18 months

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - UCL Cancer Institute, London, London
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Velindre Cancer Centre, Cardiff
  - Edinburgh Cancer Centre, Edinburgh
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Torbay Hospital, Torquay